CLINICAL TRIAL: NCT05360485
Title: Tweet4Wellness: a Social-media Based Support Group and Peer Motivation Coaches Approach to Decrease Prolonged Sitting and Increase Moderate Exercise Snacks
Brief Title: Peer Motivation Coaches, Social Media-based Support Group, and Behavior Change Strategies to Decrease Prolonged Sitting and Increase Moderate Exercise Snacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marily Ann Oppezzo, Instructor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 60388; K01HL136702 (NIH)
Record Dates: First submitted 2022-02-26; First posted 2022-05-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-03

CONDITIONS: Sedentary Behavior; Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This is preliminary efficacy, acceptability, and feasibility pilot with a randomized controlled design. The preliminary efficacy pilot will test the effects of MOV'D, a socially-supported, evidence-based behavior change technique educational and behavioral intervention to increase the number of active hours (an indirect measure of prolonged sitting bouts) (Hypothesis 1) and number of MVPA minutes (Hypothesis 2). The pilot will gather important estimates of the effect sizes, the variance, and covariance of the primary outcomes to calculate the sample size needed to power a larger trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fitbit-Only Self-Monitoring (Active Comparator): Control participants will be sent a Fitbit and study-provided account and will self-monitor physical activity for the duration of the study period (2 months).
  Interventions: Behavioral: Fitbit Self-Monitoring
- MOV'D plus Fitbit Self-Monitoring (Experimental): Treatment participants will be sent a Fitbit and study-provided account, and assigned to a private, study-created Twitter support group of 10 participants. Within the private group of 10, each participant is also further paired with a peer to be that person's peer coach, setting weekly exercise snack goals and practicing behavior change techniques.
  Interventions: Behavioral: MOV'D (Move Often eVery Day); Behavioral: Fitbit Self-Monitoring

INTERVENTIONS:
Behavioral: MOV'D (Move Often eVery Day) — The MOV'D intervention is a remotely-delivered, peer-supported intervention that delivers exercise snack (2-5 minutes of moderate to vigorous activity) and behavior change technique (BCT) videos to a private social media support group with the goal of interrupting prolonged sitting at work with MVPA minutes.
  Arms: MOV'D plus Fitbit Self-Monitoring
Behavioral: Fitbit Self-Monitoring — All participants receive a Fitbit and are told to monitor their physical activity for the duration of the study period.

SUMMARY:
The MOV'D (Move Often eVery Day) intervention is a remotely-delivered, peer-supported intervention that delivers exercise snack (2-5 minutes of moderate to vigorous activity) and behavior change technique (BCT) videos to a private social media support group with the goal of interrupting prolonged sitting at work with MVPA minutes.

The preliminary efficacy, feasibility, and acceptability trial will test the effects of MOV'D, a socially-supported, evidence-based behavior change technique educational and behavioral intervention to increase the number of active hours (an indirect measure of prolonged sitting bouts) (Hypothesis 1) and number of MVPA minutes (Hypothesis 2). This pilot will gather important estimates of the effect sizes, the variance, and covariance of the primary outcomes to calculate the sample size needed to power a larger fully powered RCT.

DETAILED DESCRIPTION:
Prolonged sitting and inadequate moderate to vigorous intensity physical activity (MVPA) are pervasive risk factors for cardiovascular disease (CVD). Recent research has shown that some benefits of moderate to vigorous physical activity can be accrued in motivationally accessible short, 2-5 minute bouts throughout the day rather than needing to be a single, longer, continuous bout. The MOV'D intervention is a novel, remotely-delivered, social-media-based intervention to interrupt prolonged sitting with short bouts of MVPA, compared with a Fitbit-only control. The investigators will randomly assign participants to either MOV'D or a Fitbit only control for one month, with a one-month follow-up, to compare immediate and prolonged effects of treatment on number of workday hours with activity break and number of MVPA minutes.

ELIGIBILITY:
Inclusion Criteria:

* have smartphone with internet capabilities
* spend more than 55% of time sedentary at work
* English literacy
* safe to exercise, assessed by the Physical Activity Readiness Questionnaire (PAR-Q)
* full-time employee at sedentary job

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in average active workday hours at post-intervention | 5 days at baseline, 5 days after 1 month treatment
  Average hours with >2 min of MVPA (Moderate to Vigorous Physical Activity) or 250 steps between 8 AM - 7 PM per workday (of five); proxy for prolonged sitting time
Change in average workday MVPA minutes at post-intervention | 5 days at baseline, 5 days after 1 month treatment
  Average minutes of moderate to vigorous minutes, or minutes above 3 METs per workday (of five) at

SECONDARY OUTCOMES:
Change in average active workday hours at follow-up | 5 days at baseline, 5 days post 1-month follow-up
  Average hours with >2 min of MVPA or 250 steps between 8 AM - 7 PM per workday (of five); proxy for prolonged sitting time
Change in average workday MVPA minutes at follow-up | 5 days at baseline, 5 days post 1-month follow-up
  Average minutes of moderate to vigorous minutes, or minutes above 3 METs +per workday (of five)

CONTACTS AND LOCATIONS:
Overall Officials: Marily A. Oppezzo, PhD MS, RDN, DipACLM, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be shared upon request

REFERENCES:
- [Derived] Monteiro A, Moore J, Aikens R, Duckworth A, Gross JJ, Schwartz D, Baiocchi M, Prochaska JJ, Oppezzo M. A Work-Based, Fully Remote, and Peer-Supported Exercise Snack Behavior Change Intervention (MOV'D): Protocol for a Randomized Controlled Pilot Trial. JMIR Res Protoc. 2025 Aug 7;14:e64455. doi: 10.2196/64455. PMID 40773742
- [Derived] Zamora AN, Zeitlin AB, Moore JB, Oppezzo M. Exploring Perceptions, Barriers, and Facilitators of Participation in an Exercise Snack Intervention Among U.S. Office Workers: Findings From a Pilot Study. Am J Health Promot. 2025 May 4:8901171251338217. doi: 10.1177/08901171251338217. Online ahead of print. PMID 40320694